CLINICAL TRIAL: NCT03199547
Title: Pre-delivery Administration of Azithromycin to Prevent Neonatal Sepsis and Death: a Phase III Double-blind Randomized Clinical Trial
Brief Title: Pre-delivery Administration of Azithromycin to Prevent Neonatal Sepsis & Death
Acronym: PregnAnZI-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SCC 1532
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Neonatal SEPSIS
MeSH Terms: conditions — Neonatal Sepsis | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: This is a Phase III, double-blind, placebo controlled randomized clinical trial. Women attending the study health facilities in labour will be randomized to receive either a single dose of oral AZI (2g) or placebo (1:1)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The active study drug and placebo will look identical and will not be identifiable. The study drugs will be allocated to the participants according to the randomisation number
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZITHROMYCIN (Experimental): A single dose of 2G Azithromycin or Placebo will be administered orally to women in labour
  Interventions: Drug: Azithromycin
- Placebo oral tablet (Placebo Comparator): A single dose of 2G Azithromycin or Placebo will be administered orally to women in labour
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Azithromycin — The women will be randomized to receive a single dose of Azithromycin or Placebo
  Arms: AZITHROMYCIN
Drug: Placebo Oral Tablet — The women will be randomized to receive a single dose of Azithromycin or Placebo
  Arms: Placebo oral tablet

SUMMARY:
Though maternal and neonatal health are high priority areas for international development, maternal and neonatal mortality remain unacceptably high. Worldwide there are 1 million maternal and 4 million neonatal deaths every year and half of them occur in sub-Saharan Africa.

Post-partum and neonatal severe bacterial infections, namely sepsis, are leading causes of maternal and neonatal deaths in sub-Saharan Africa. Newborns can be infected during labour - when passing through the birth canal - and also during the first days/weeks of life, as a consequence of the close physical contact with the mother, when the latter carriers bacteria. As the mother is an important source of bacterial transmission to the newborn, treating mothers with antibiotics during labour should decrease their bacterial carriage and therefore lower transmission to the newborn. As carriage is a necessary step towards severe disease, this intervention should in turn result in the lower occurrence of severe bacterial disease and mortality during the neonatal period.

In many high-income countries, pregnant women are screened during pregnancy for vaginal carriage of Group B Streptococcus, the bacteria responsible for the vast majority of neonatal sepsis in the developed world. If women are carriers, they are treated with intravenous antibiotics during labour to decrease the risk of severe disease to their off-spring. Although this intervention has been successful in developed countries, infrastructure and resource limitations in regions like sub-Saharan Africa prevent both screening and use of intravenous antibiotics. Also, in Africa several bacterial pathogens are responsible for neonatal sepsis and the antibiotics needed in the continent should cover a wider number of bacteria; and ideally cover also bacteria responsible for severe post-partum disease in the mother.

We will conduct a large trial in West Africa, The Gambia and Burkina Faso, with the main objective of determining if a single dose of an oral antibiotic given to women during labour decreases newborn mortality. The trial will also assess the effect of the antibiotic on lowering newborns and maternal hospitalization during the first week's post-partum. We have selected an antibiotic (azithromycin) that in sub-Saharan Africa has already been used for elimination of other prevalent diseases such as trachoma. This antibiotic is safe, requires a single oral administration, has no special storage requirements and has the potential to eliminate most of the bacteria commonly causing severe disease in newborns and post-partum women in the continent. Very important this antibiotic is not widely used in clinical care in the continent, and therefore, any temporal increase of resistance induced by the intervention should not have implications on current treatment guidelines.

Before going to the large trial proposed here (12,000 women to be recruited), we have generated robust preliminary data on the effect of the intervention in a proof-of-concept trial conducted in The Gambia (829 women and their offspring recruited). We found that in fact, babies born from mothers who had taken this antibiotic during labour were less likely to carry bacteria that can potentially cause severe disease. These babies were also three times less likely to have bacterial skin infections or umbilical infections, both highly common among African newborns. Besides, fever or mastitis (again both very common in the region) during the post-partum period were four times lower among mothers who had taken the antibiotic during labour. Such trial confirmed our hypothesis of impact on bacterial transmission but it was too small to assess the effect of the antibiotic on mortality and hospitalizations. The preliminary trial also showed that women from the azithromycin group were less likely to need antibiotics for treatment infections during the puerperal period, decreasing then the pressure on the scarcity of antibiotics available in the continent.

The advantages of our approach are its simplicity, low cost and the possibility of protecting both mothers and babies with the same intervention.

DETAILED DESCRIPTION:
other data elements, such as eligibility criteria or outcome measures. (Limit: 32,000 characters) Project title: Pre-delivery administration of azithromycin to prevent neonatal sepsis and death: a phase III double-blind randomized clinical trial Acronym: PregnAnZI-2

LIST OF INVESTIGATORS

Chief Investigator:

Dr Anna Roca, PhD MRC Unit The Gambia PO Box 273 Banjul The Gambia, West Africa aroca@mrc.gm

Co-Investigators:

Prof Umberto D'Alessandro Director - MRC Unit The Gambia PO Box 273 Banjul The Gambia, West Africa udalessandro@mrc.gm

Dr Christian Bottomley PhD Trial Statistician London School of Hygiene and Tropical Medicine London Christian.bottomley@lshtm.ac.uk

Dr Halidou Tinto PhD Site PI Burkina Faso Clinical Research Unit of Nanoro Burkina Faso tintohalidou@yahoo.fr

Clinical Trial Coordinators:

Dr Bully Camara MD MRC Unit The Gambia PO Box 273 Banjul The Gambia, West Africa +2204495917

Dr Marc Tahita Clinical Research Unit of Nanoro Burkina Faso BACKGROUND AND RATIONALE Neonatal and maternal sepsis are major contributors to the high burden of mortality in sub-Saharan Africa (SSA). Bacterial infections are leading causes of neonatal deaths, representing 1 out of 3 deaths in this age group (1).

Neonatal sepsis is the consequence of bacterial infection during early life. Newborns may be infected during labour (through the birth canal) or during the first days/weeks of life, when they may become infected because of the close physical contact with the mother, if the latter carries bacteria (i.e. in the nasopharyngeal tract), a common occurrence in resource-limited settings, particularly in SSA. Streptococcus pneumoniae and group A Streptococcus are important in the late neonatal period (from the second week of life), while group B Streptococcus (GBS), Staphylococcus aureus and Escherichia coli occur often in both the early and late neonatal periods (2).

AZI is a semi-synthetic azalide macrolide that is structurally related to erythromycin but has a broader spectrum of antibacterial activity, improved tissue penetration and a more favourable pharmacokinetic profile (3). Azithromycin is a cheap, wide spectrum, oral antibiotic that is safe to use in mothers and newborns, does not require special storage conditions, and can be delivered at the most peripheral level of care.

Between 2013 and 2015, we conducted as first proof-of-concept, a double-blind randomized trial on the effect of 2g of AZI administered to Gambian women in labour on maternal and neonatal bacterial carriage (4). The primary endpoint was bacterial carriage at day 6 in the newborn (i.e. S.aureus, GBS or S.pneumoniae). The rationale for the study was that this intervention would decrease bacterial carriage of the study bacteria both, in the mother and the newborn and consequently the risk of invasive bacterial disease or sepsis. We found that the intervention substantially reduced the prevalence of carriage of each of these three bacteria, both in the newborn and the mother, during the entire neonatal/puerperal period (4).

Figure 1. Prevalence of nasopharyngeal bacterial carriage during the neonatal period.

(a) Newborn (b) Mother1

1 Maternal nasopharyngeal swab at day 0: collected before the intervention was given.

Our study also showed that women in the AZI group had a lower prevalence of the study bacteria in the breast milk during the entire neonatal period (day 6: 9.6% vs 21.9%, RR=0.44, p<0.001) and in the vaginal tract (8-10 days: 13.2% vs 24.2% RR=0.55 - p<0.001).

Although the study was not designed to evaluate clinical endpoints, prevalence of these endpoints decreased significantly in the AZI group (5). The use of antibiotics, and the occurrence of fever, mastitis and puerperal infections were significantly lower in the AZI group (Table 1). Newborns in the intervention group had fewer infections (skin infections, umbilical infections, ear infections, conjunctivitis or mild sepsis) during the neonatal period (Table 2). There were also fewer neonatal deaths due to severe infections in the AZI group (0.4% versus 1.4% excluding neonates with severe congenital malformations).

Table 1. Clinical endpoints and antibiotic use of study women during the puerperal period.

MATERNAL Azithromycin (N=414) Placebo (N=415) RR(95%CI) p-value Maternal infections n(%) n(%) Mastitis 6(1.4) 21(5.1) 0.29(0.12,0.70) 0.005 Puerperal sepsis 4(1.0) 5(1.2) 0.80(0.22,2.97) 1 Related infections 3(0.7) 9(2.2) 0.33(0.09,1.23) 0.143 Others 2(0.5) 5(1.2) 0.40(0.08,2.06) 0.451 Any of above 17(4.1) 38(9.2) 0.45(0.26,0.78) 0.005 Fever 8(1.9) 24(5.8) 0.33(0.15,0.74) 0.006 Use of antibiotic (for clinical care) 25(6.0) 42 (10.1) 0.58(0.36,0.94) 0.031 Table 2. Clinical endpoints and antibiotic use of study children during the neonatal period.

NEONATES Azithromycin (N=419) Placebo (N=424) RR(95%C) p-value Neonatal infections n(%) n(%) Skin infection 13(3.1) 27(6.4) 0.49(0.25,0.93) 0.034 Umbilical infection 1(0.2) 4(0.9) 0.25(0.03,2.25) 0.374 Conjunctivitis 37(8.8) 45(10.6) 0.83(0.55,1.26) 0.417 Otitis 3(0.7) 5(1.2) 0.61(0.15,2.52) 0.725 Oral infection 12(2.9) 13(3.1) 0.93(0.43,2.02) 1 Sepsis 18(4.3) 15(3.5) 1.21(0.62,2.38) 0.598 Meningitis 0(0.0) 1(0.2) NA 1 Pneumonia 3(0.7) 4(0.9) 0.76(0.17,3.37) 1 Any of above 76(18.1) 101(23.8) 0.76(0.58,0.99) 0.052 Fever 54(12.9) 43(10.1) 1.27(0.87,1.85) 0.235 Use of any antibiotic (for clinical care) 43(10.1) 42(10.0) 0.99(0.66,1.5) 1 The time point when the endpoints occurred during the follow-up period are summarized in Figure 2 below.

Figure 2. Proportion of mothers and newborns infected at different points during the follow up.

p-values from the log-rank test (mothers p=0.001, newborns p=0.04) AZI was safe for both the mothers and the newborns. Hypertrophic pyloric stenosis (HPS) was not observed in any of the study children during the 2-month follow up period (4).

Azithromycin is a cheap, wide spectrum, oral antibiotic that is safe to use in mothers and newborns, does not require special storage conditions, and can be delivered at the most peripheral level of care.

In the trial presented here, we want to assess the impact of using AZI during labour on neonatal mortality as well as maternal and neonatal sepsis and infant growth. If successful, this simple intervention could be easily implemented through the health system at the most peripheral level of care. It has the potential to achieve wide coverage in SSA where low-cost interventions aiming at reducing neonatal mortality are urgently needed. In addition, the intervention should concomitantly protect women and newborns. Azithromycin resistance will also be monitored as the former trial showed high rates of AZI resistance for S. aureus. However, AZI is not widely used in SSA for clinical treatment and therefore any short-term resistance arising from the intervention would have little impact on clinical care.

References

1. Lawn JE, Cousens S, Zupan J et al. (2005) 4 million neonatal deaths: When? Where? Why? Lancet 365: 891-900. S0140-6736(05)71048-5.
2. Sigauque B, Roca A, Mandomando I et al (2009) Community-acquired bacteremia among children admitted to a rural hospital in Mozambique. Pediatr Infect Dis J 28: 108-113.
3. Chico RM, Chandramohan D (2011) Azithromycin plus chloroquine: combination therapy for protection against malaria and sexually transmitted infections in pregnancy. Expert Opin Drug Metab Toxicol 7: 1153-1167.
4. Roca A, Oluwalana C, Bojang A et al (2016). Oral azithromycin given during labour decreases bacterial carriage in the mother and their offspring: a double-blind randomized trial. Clin Microbiol Infect. Jun;22(6):565.
5. Oluwalana C, Camara B, Bottomley C, et al (2017). Azithromycin in labor lowers clinical infections in mothers and newborns: a double-blind trial. Pediatrics; 139(2).

   TRIAL DESIGN

   This is a multi-country phase III, double-blind, placebo-controlled, randomised trial in which 12,500 women in labour will be randomised to receive either a single dose of 2g of oral azithromycin or placebo (ratio 1:1). Pregnant women (age ≥16 years) will be identified during antenatal clinic visits in several health facilities in The Gambia and Burkina Faso; and will be asked to provide written informed consent. Recruitment will take place when these women attend the study health facilities in labour.

   INCLUSION AND EXCLUSION CRITERIA Pregnant women (age ≥16 years) will be identified during antenatal clinic visits and asked to provide written informed consent. During labour they will be screened and recruited unless they have any of the following exclusion criteria: planned caesarean section, ante-partum haemorrhage, known allergy to macrolides, confirmed intrauterine death or a known severe congenital malformation. The randomisation number will only be assigned after the screening.

   TRIAL OBJECTIVES

   The primary objective of the study is to assess the effect of one oral dose of AZI (2g) given to women in labour on neonatal sepsis and mortality (from birth to 28 days). Deaths due to severe birth asphyxia (Apgar score <3 at 1 min); severe congenital malformations and very low birth weight (VLBW) (<1.5Kg) will be excluded. Note: Those deaths excluded from the primary objective are considered in some of the secondary objectives below.

   Secondary objectives of the trial include the effect of the intervention on other clinical endpoints (for both neonates and mothers) and on microbiological endpoints (prevalence of carriage and resistance of different bacterial pathogens):

   (i) Neonates

   a. Efficacy on clinical neonatal sepsis b. Efficacy on neonatal deaths, excluding those due to severe birth asphyxia, severe congenital malformations or VLBW c. Efficacy on severe birth asphyxia and associated deaths d. Efficacy on culture-confirmed neonatal sepsis e. Efficacy on all cause-hospitalisation during the follow-up period (during the first 28 days) f. Efficacy on sepsis and all cause mortality among VLBW g. Efficacy on skin infection h. Efficacy on bacterial conjunctivitis i. Efficacy on umbilical cord infections j. Efficacy on clinical malaria k. Efficacy in the use of antibiotics during the neonatal period

   (ii) Infants (Children of the first 1,000 mothers recruited per country followed-up to 1 year)
   1. Efficacy on all cause-mortality
   2. Efficacy on malnutrition - Height-for-age (HAZ), weight-for-age (WAZ), weight-for-height (WHZ), body mass index-for-age, head circumference-for-age, and MUAC for age (28 days; 6 and 12 months)

   (iii) Mothers (up to 28 days) a. Efficacy on post-partum sepsis b. Efficacy on post-partum mastitis c. Efficacy on post-partum malaria d. Efficacy on post-partum fever e. Efficacy on use of post-partum antibiotics f. Efficacy on all post-partum hospitalisations g. Efficacy on all post-partum mortality (iv) Microbiological objectives (for hospitalised newborns)
   1. Efficacy on prevalence of S. pneumoniae and Klebsiella spp in the nasopharynx
   2. Efficacy on prevalence of E.coli and Pseudomonas spp in rectal swabs (RS)
   3. Efficacy on prevalence of S. aureus, GBS, GAS in the oropharyngeal swabs

   (v) Microbiological objectives (random selection of 250 participant pairs in each country)
   1. Efficacy on prevalence of S. pneumoniae and Klebsiella spp in the nasopharynx of study infants at different time points.
   2. Efficacy on prevalence of E. Coli, Klebsiella spp and Pseudomonas spp from RS collected from infants at different time points.
   3. Efficacy on prevalence of S. aureus, GBS and GAS in the oropharynx of infants at different time points.
   4. Efficacy on prevalence of S. aureus, GBS, GAS, E. coli, Pseudomonas spp and Klebsiella in the breast milk of the study women at different time points.
   5. Efficacy on prevalence of S. pneumoniae and Klebsiella spp in the nasopharynx of study women one week after the intervention.
   6. Efficacy on the prevalence of S. aureus, GBS and GAS in the oropharynx of study women one week after the intervention.
   7. Effect of the intervention onAZI, oxacillin and amoxicillin resistance among isolates of S. aureus, GBS, GAS, S. pneumoniae, Klebsiella spp, E. coli and Pseudomonasspp at different time points during the follow-up period.

   (vi) Clinico-microbiological sub-analysis (sub-group of approximately 4,000 for whom pre-intervention recto-vaginal swab is collected during labour)

   a. Efficacy of the intervention on neonataland maternal outcomes [see (i) and (iii)] when women are carrying S. aureus, Klebsiella spp, Pseudomonas spp, GBS, GAS or E. coli in the recto-vaginal tract.

   Tolerability of AZI given during labour will be monitored for all recruited women.

   Other aspects of the study such as Qualitative research and Health economics are not included in the clinical trial protocol but a summary of the objectives are as follows:

   (vii) Qualitative research: a. Perceptions and acceptability by pregnant women and the study communities on the taking antibiotic during labour.

   (viii) Health economics

   a. Costs of delivering AZI during labour in a health facility. b. Cost of a newborn death. c. Hospitalisation treatment costs. d. Disability Adjusted Life Year averted from delivering the intervention. PARTICIPANTS AND SAMPLES We will recruit 12,500 women and their newborns. Approximately half of this number of women will be recruited in The Gambia and half in Burkina Faso. However, the recruitment will be competitive and if one country does not reach the numbers within the time period expected, the other will increase the recruitments.

   Figure 3. Length of follow-up of study participants and visits.

   *Visit at Day 0/1 (recruitment at the health facility and discharge from the health facility) and visit at Day 28 is the same for all the study participants. The additional active visits are only for participants included in one of the sub-studies.

   All study participants will be followed for 28 days. During this follow-up period, samples will be collected if they are hospitalized with suspicion of sepsis (mothers and newborns). Clinical samples to conduct sepsis work up will be collected. For newborns hospitalized with clinical suspicion of sepsis, we will also collect nasopharyngeal swabs (NPS), oropharyngeal swabs (OPS) and rectal swabs (RS).

   For 250 participant pairs recruited in the carriage sub-study. Samples will be collected according to the table below.

   Table 3. Samples collected from the participants included in the carriage sub-study.

   Day 01 Day 6 (±2 days) Day 28 (±4 days) 4 Months (±2 weeks) Mother Recto-Vaginal swab X2 Nasopharyngeal swab X2 X Oropharyngeal swab X2 X Breast Milk X X X Newborn Nasopharyngeal swab X3 X X X Oropharyngeal swabs X3 X X X Rectal swabs X3 X X X 1Samples at day 0 will be collected at the health facilities. 2For the women, samples will be collected before treatment; 3Within 4 hours after birth.

   For infants of the first 1,000 mothers s participating in the anthropometrical sub-study. These children will be followed for 1 year but no additional samples will be collected. Anthropometric information will be collected during the additional visits at 6, 9 and 12 months; and information of AE will be collected.

   CENTRES INVOLVED IN THE TRIAL

   In The Gambia, we will conduct the trial at Bundung Maternal and Child Health Hospital and Serrekunda Health Facility. Bundung Maternal and Child Health Hospital is where the proof-of-concept trial was conducted. The hospital delivers approximately 5,000 babies each year and is located on the Gambian coast, 15 km from the MRC The Gambia headquarters. Pregnant women usually have 2-3 antenatal visits during the second and third trimester and they are kept in the health centre for approximately 6 hours after delivery. Serrekunda Health Facility is located approximately 15Km from both the Bundung Maternal and Child Health Hospital and the MRC The Gambia headquarters. Approximately, 2,000 deliveries take place per year. In The Gambia, maternal mortality ratio is 461 deaths/100,000 live births (4) and infant mortality rate is above 50 deaths/1,000 live births (5).

   In Burkina Faso, the study will be carried out at the Clinical Research Unit of Nanoro (CRUN) located in the rural central west region of the country. In 2013, the total population of the Nanoro Health district was estimated at 158,127 people. There are 14 peripheral health facilities (covering 70 villages) around the referral hospital, all with maternity and extended program of immunizations (EPI) services. Seven to 10 of these health facilities will be part of the trial. The epidemiological profile of diseases remains dominated by communicable infectious diseases. Maternal mortality rate is 300 deaths/100,000 live births and infant mortality rate is 78.3 deaths/1,000 live births. A Health and Demographic Surveillance System (HDSS), which covers a total population of about 60,000 people in 24 villages (7 health facilities) was set up in 2009 by the CRUN within the Health district catchment area.

   ALLOCATION OF PARTICIPANTS Randomisation lists based on permuted blocks will be created independently for each country, and blister packs will be numbered according to the list. The trial will comply with Good Clinical Practices (GCP).

   RISK TO THE SAFETY OF THE TRIAL
   1. Hyperpyloric stenosis (HPS). Azithromycin is associated with HPS in infants (6) although it is uncertain in the context of azithromycin treated breast feeding women (7). Typically, infants with HPS do not show any symptoms at birth but they develop projectile vomiting and other metabolic abnormalities during the first few weeks of life. Data generated in our pilot study showed that azithromycin reaches the breast milk and traces are still detectable in samples collected at day 28 (8). There is some evidence that HPS is less frequent in SSA (9). In our pilot study none of the 419 children whose mother received azithromycin developed HPS (8). Nevertheless, newborns will be carefully followed up for signs of HPS.
   2. Azithromycin resistance. Azithromycin is not routinely used for clinical care in SSA and has a wide antimicrobial spectrum (10). For these reasons it has been used in several successful mass drug administration (MDA) campaigns, including trachoma and yaws control and elimination (11;12), and in clinical trials for the prevention of malaria in pregnancy and preterm births (13). Most studies have shown to varying degrees that resistant bacteria can be selected after a single dose. Nevertheless, in the absence of antibiotic pressure, resistance disappears due to the lower fitness of resistant bacteria (14). Studies that have used azithromycin for MDA, in which thousands of people were treated at the same time, have shown that S.pneumoniae resistance is only maintained for more than a few months in communities where the baseline prevalence of resistance is high (15). In The Gambia azithromycin resistance after MDA for trachoma elimination reverted to baseline levels 6 months after the intervention (16). In our pilot study, resistance of S.aureus was high 28 days after treatment but decreased to baseline levels 12 months after treatment (Bojang et al in prep). As azithromycin is not used in standard clinical care, there would be little selective pressure on resistant bacteria. In addition, it is interesting to note that in our pilot trial women in the azithromycin group used other antibiotics less often than women in the placebo arm (2). This suggests that the intervention might decrease selective pressure on the few antibiotics available for standard clinical care in the region. Resistance to azithromycin and other antibiotics among the trial participants will be assessed in the proposed study.

   SAMPLE SIZE CALCULATION In our proof-of-concept trial, the prevalence of bacterial carriage in the azithromycin group decreased by more than 50%, and there were 6 neonatal deaths (1.4%) (primary endpoint as defined above) in the placebo arm compared to 2 (0.4%) in the azithromycin arm (70% reduction).

   We assume that mortality in the placebo arm will be at least 1.4% - this is a conservative estimate as in the proof-of-concept trial neonates were closely followed up during the first week of life and this probably decreased the risk of death. Assuming the intervention reduces neonatal mortality by 40%, we would need 5,800 women per arm to show a significant difference at 80% power and 5% significance level. And allowing for 8% loss to follow-up, we would need to recruit a total of 12,500 women.

   Up to two thirds of these women will be recruited in the Gambia, and the remainder will be recruited in Burkina Faso, depending on the pace of recruitment in both countries. Maternal and infant mortality rates in these two countries are similar. The sample size would also provide reasonable power for the secondary endpoints of maternal and neonatal infection, hospitalisation and antibiotic use, since their occurrence is higher than neonatal death.

   As during the trial we have observed a mortality of approxiamtely half of the expected, we have modified the endpoint to a composite endpoint of mortality or sepsis. This composite endpoint prevalence is approximately 2.1% of the total sample size. Assuming the intervention reduces the endpoint by 28%, 12,000 participants gives us 80% power at a 5% significance level to detect differences by study arm.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women in labour (aged 16 years or more) attending the study health facilities for delivery who have previously given consent and willing to continue participation

Exclusion Criteria:

Known HIV infection. Any chronic or acute conditions of the women that might interfere with the study as judged by the research clinician.

Planned travelling out of the catchment area during the following 28 days Planned caesarean section or known required referral Known severe congenital malformation Intrauterine death confirmed before randomisation Known allergy to macrolides Already participating in another trial

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women attending study health facilities for delivery will be enrolled
Enrollment: 11985 (Actual)
Dates: Start 2017-10-21 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
neonatal sepsis and mortality | from Birth to Day 28
  The primary endpoint of the study is a composite endpoint of prevalence of neonatal sepsis and mortality rate (from birth to 28 days) (deaths from severe birth asphyxias, major congenital malformations and VLBW are excluded from the primary endpoint).

SECONDARY OUTCOMES:
Neonatal sepsis-Early-onset of Culture confirmed sepsis | Day 1- Day 3
  isolation of a miro-organism that is not a common contaminant from a normally sterile body site (i.e. blood or CSF)
Early-onset clinical sepsis | Day 1- Day 3
  neonate hospitalised within 3 days of life and who in the absence of another recognisable congenital infection had at least one laboratory criteria and either: respiratory distress (one criterion required) or at least two clinical criteria
Late-onset culture confirmed sepsis | Day 3 - Day 28
  isolation of a micro-organism that is not a common contaminant from a normally sterile body (i.e. blood or CSF) site if a microorganism has been observed in the gram stain (i.e. CSF)
Late-onset clinical sepsis | Day 3- Day 28
  neonate hospitalised with at least one laboratory criteria and either: respiratory distress (twocriteria required), OR one feature of respiratory distress and one other clinical criterion OR at least two other clinical criteria
All-caused hospitalisation during the follow up period | 28 days forAll study participants will be followed for 28 days except those participating in the sub-studies; 4 months for children in carriage sub-study; 12 months for children participating in the anthropometrical sub-stud
  Hospitalisation will be defined as admission to an inpatient ward or at least a 12 hour stay. We will exclude from this endpoint all hospitalizations due to injuries
Infant mortality | Birth to 12 Months
  All-cause mortality excluding injuries (only for those included in the anthropometrical sub-study).
Malnutrition and Severe malnutrition | At 6, 9 and 12 months of age
  through anthropometrical measurements and using WHO child-growth standards to calculate Z-scores for height-for-age (HAZ), weight-for-age (WAZ), weight-for-height (WHZ), head circumference-for-age, and MUAC for age [WHO Anthro version 3.2.2, January 2011]. Children with z-scores <-2SD and <-3SD will be classified as malnourished and severely-malnourished, respectively
Post-partum sepsis- Women | Day 1 to Day 28
  this will be defined as admission of the mother for endometritis (defined below) or culture-confirmed infection of sterile site (i.e. blood of CSF; or bacteria detected in the gram stain) or wound infection (see definition below) [23].
  * Endeometritis: at least two of the following signs of uterine tenderness, fever (>38.0 oC), foul-smelling or purulent lochia, or vaginal discharge diagnosed by clinicians and/or nurses.
  * Wound infection is defined as perineal wound infection among vaginal parturients or cesarian wound infection among ceasarean section parturients
All-cause maternal hospitalisation | Day 1 to day 28
  Hospitalisation will be defined as admission to an inpatient department or a visit to an emergency department that results in at least a 12-hour stay excluding hospitalizations due to injuries

CONTACTS AND LOCATIONS:
Overall Officials: Anna Roca, PhD, Principal Investigator — MRC Unit The Gambia
Locations (2):
- Clinical Research Unit of Nanoro, Nanoro, Burkina Faso
- Medical Research Council Unit The Gambia, Banjul, The Gambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bojang A, Chung M, Camara B, Jagne I, Guerillot R, Ndure E, Howden BP, Roca A, Ghedin E. Genomic approach to determine sources of neonatal Staphylococcus aureus infection from carriage in the Gambia. BMC Infect Dis. 2024 Sep 9;24(1):941. doi: 10.1186/s12879-024-09837-5. PMID 39252007
- [Derived] Getanda P, Jagne I, Bognini JD, Camara B, Sanyang B, Darboe S, Sambou E, Barry M, Kassibo K, Cham A, Mendy H, Singateh BKJ, Ndure E, Rouamba T, Bojang A, Bottomley C, Howden BP, D'Alessandro U, Tinto H, Roca A; PregnAnZI-2 Carriage Study Group. Impact of Intrapartum Azithromycin on the Carriage and Antibiotic Resistance of Escherichia coli and Klebsiella pneumoniae in Mothers and Their Newborns: A Substudy of a Randomized, Double-Blind Trial Conducted in The Gambia and Burkina Faso. Clin Infect Dis. 2024 Dec 17;79(6):1338-1345. doi: 10.1093/cid/ciae280. PMID 38752311
- [Derived] Roca A, Camara B, Bognini JD, Nakakana UN, Some AM, Beloum N, Rouamba T, Sillah F, Danso M, Jones JC, Graves S, Jagne I, Getanda P, Darboe S, Tahita MC, Ndure E, Franck HS, Edmond SY, Dondeh BL, Nassa WGJ, Garba Z, Bojang A, Njie Y, Bottomley C, Tinto H, D'Alessandro U; PregnAnZI-2 Working Group. Effect of Intrapartum Azithromycin vs Placebo on Neonatal Sepsis and Death: A Randomized Clinical Trial. JAMA. 2023 Mar 7;329(9):716-724. doi: 10.1001/jama.2022.24388. PMID 36881034

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT03199547/SAP_000.pdf